CLINICAL TRIAL: NCT03931434
Title: Effect of Aged Garlic Extract (AGE) on Progression of Coronary Atherosclerosis in Persons With Type 2 Diabetes Mellitus
Brief Title: Effect of Aged Garlic Extract (AGE) on Improving Coronary Atherosclerosis in People With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Matthew J. Budoff, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Garlic-5
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Coronary Arteriosclerosis; Endothelial Dysfunction; Type 2 Diabetes Mellitus
Keywords: coronary artery disease; Endothelium
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Double Blind Placebo Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aged Garlic Extract (AGE) (Active Comparator): 2400mg of Aged Garlic Extract (AGE)
  Interventions: Dietary Supplement: Aged Garlic Extract (AGE)
- Placebo (Placebo Comparator): The Placebo does not contain any Aged Garlic Extract (AGE)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Aged Garlic Extract (AGE) — 2400mg of Aged Garlic Extract (AGE)
  Arms: Aged Garlic Extract (AGE)
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this research study is to see the effect of taking Aged Garlic Extract (AGE) on the progression of coronary plaque, a condition called atherosclerosis, in people diagnosed with Diabetes.

DETAILED DESCRIPTION:
This clinical trial is to determine on progression rates of low attenuation plaque under influence of Aged Garlic Extract as compared to placebo over the 1year period in individuals with Type 2 Diabetes Mellitus.The study also examines the effect of Aged Garlic Extract on endothelial function and arterial stiffness which was measured by cardio-ankle vascular index (CAVI) over the 3months period.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-75 years
* Known Diabetes Mellitus (HgA1c >6.5%, fasting blood sugar >125 mg/dl, taking anti- diabetes medications)
* Subjects must provide written informed consent after the scope and nature of the investigation has been explained to them
* Calcium Score >20 at baseline

Exclusion Criteria:

* A contraindication to AGE including: known hypersensitivity to drug.
* Any unstable medical, psychiatric or substance abuse disorder that in the opinion of the investigator or principal investigator is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study
* Weight in excess of 350 pounds
* Bleeding disorder
* History of known coronary artery disease, myocardial infarction, stroke or life- threatening arrhythmia within the prior six months
* NYHA Class II- IV heart failure
* History of malignancy within the last 5 years (other than skin cancer) or evidence of active cancer which would require concomitant cancer chemotherapy
* Serum creatinine > 1.4 mg/dl
* Triglycerides > 400 at visit 1
* Drug or alcohol abuse, or current intake of more than 14 standard drinks per week
* Concurrent enrollment in another placebo-controlled trial
* Partial ileal bypass or known gastrointestinal disease limiting drug absorption
* Current tobacco use
* Current use of anticoagulants (except for anti-platelet agents)
* Renal failure
* History of hypertensive encephalopathy or cerebrovascular accident
* Hematological or biochemical values at screening outside the reference ranges considered as clinically significant in the opinion of the investigator or PI
* Pregnancy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Progression rates of low attenuation plaque under influence of Aged Garlic Extract (AGE) as compared to placebo. | 12 months
  Progression rates of low attenuation plaque under influence of Aged Garlic Extract (AGE) as compared to placebo.

SECONDARY OUTCOMES:
Rate of change in inflammatory biomarkers (CRP,IL-6) | 12 months
  Rate of change in inflammatory biomarkers
Rate of change in endothelial function | 3 months and 12 months
  Endothelial Function and arterial stiffness measured by cardio-ankle vascular index (CAVI)

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles Biomedical Research Institute at Harbor UCLA Medical Center, Torrance, California, United States